CLINICAL TRIAL: NCT00005949
Title: Phase II Study of Melanoma Vaccine (NSC #683472/675756, IND #6123) and Low-Dose, Subcutaneous Interleukin-2 in Advanced Melanoma
Brief Title: Vaccine Plus Interleukin-2 in Treating Patients With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02337; CLB-509901; U10CA031946 (NIH); CDR0000067886 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interleukin-2; Protein Subunit Vaccines

ARMS (1):
- Treatment (gp100:209-217, aldesleukin ) (Experimental): Patients receive gp100:209-217(210M) emulsified in Montanide ISA-51 SC on day 1 and interleukin-2 SC on days 1-5 and 8-13. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression. Patients with a CR receive 3 additional courses after achieving CR.
  Interventions: Biological: aldesleukin; Biological: gp100:209-217(210M) peptide vaccine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Biological: gp100:209-217(210M) peptide vaccine — Given SC
  Other Names: G9 209-2M; gp100:209-217(210M)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of vaccine therapy plus interleukin-2 in treating patients who have advanced melanoma. Vaccines made from a person's cancer cells may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Melanoma vaccine plus interleukin-2 may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine clinical response rates in patients with advanced melanoma treated with gp100:209-217(210M) melanoma vaccine and low-dose interleukin-2.

II. Assess response duration and progression-free intervals in these patients receiving this treatment.

OUTLINE:

Patients receive gp100:209-217(210M) emulsified in Montanide ISA-51 subcutaneously (SC) on day 1 and interleukin-2 SC on days 1-5 and 8-13. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression. Patients with a complete response (CR) receive 3 additional courses after achieving CR.

Patients are followed every 9 weeks for 3 years or until disease recurrence.

PROJECTED ACCRUAL: A total of 25-50 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed cutaneous melanoma with clinical evidence of distant, metastatic, unresectable regional lymphatic, or extensive in-transit recurrent disease
* HLA-A2*0201 positive by genotyping
* Measurable disease as defined by the following:

  * At least 1 lesion accurately measured in at least 1 dimension
  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
  * Lesions considered intrinsically nonmeasurable include:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
    * Lesions situated in a previously irradiated area
* No ocular or mucosal melanoma
* No prior or concurrent liver or brain metastases
* Performance status - ECOG 0-1
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL
* LDH normal
* Bilirubin normal
* AST no greater than 2.5 times upper limit of normal
* Creatinine normal
* No congestive heart failure, angina, or symptomatic cardiac arrhythmia
* No myocardial infarction within the past 6 months
* No severe chronic pulmonary disease
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No primary or secondary immunodeficiency or autoimmune disease
* No currently active second malignancy (e.g., patient has completed therapy and is considered unlikely to have recurrence within 1 year) other than nonmelanoma skin cancer
* At least 4 weeks since prior immunotherapy
* No prior interleukin-2
* No prior whole cell or gp100:209-217(210M)-targeted melanoma vaccine
* No other concurrent cytokines or growth factors
* At least 4 weeks since prior chemotherapy
* At least 1 month since prior systemic corticosteroids
* No concurrent systemic, inhaled, or topical corticosteroids
* At least 1 month since other prior immunosuppressive medication
* No antihypertensive medications from 1 day prior until 2 days after first course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-03; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Clinical response rate (CR or PR) | From the start of treatment until disease progression/recurrence, assessed up to 3 years

SECONDARY OUTCOMES:
Response duration | Up to 3 years
  The Kaplan-Meier method will be used to estimate duration of response.
Progression-free intervals | Up to 3 years
  The Kaplan-Meier method will be used to estimate time to progression.
Immunologic response rate using ELISPOT assay | Up to 3 years
  Described in terms of frequency and kinetics. Agreement between clinical and immunological response will be measured using the kappa coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: John Roberts, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States